CLINICAL TRIAL: NCT05088031
Title: Shock Wave Therapy Versus Mechanical Traction on Mechanical Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Merit University (Other)
Responsible Party: Principal Investigator, Ahmed Assem, Lecturer of Physical Therapy, Merit University
Other Study IDs: Mechanical LBP
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1- Group ( A): 20 patients underwent shock wave therapy: 1-Group (A): 20 patients would undergo shock waves plus traditional physical therapy. One thousand shock waves (7 times per sec) were applied at 2.5 Hz at low energy flux densities of 0.01-0.16 mJ/mm2 using a 17 mm head for 15 minutes on alternate days for four weeks for a total of 12 sessions14.
  Interventions: Device: shock waves therapy
- 2-Group (B): 20 patients would undergo intermittent mechanical traction: 2-Group (B): 20 patients would undergo intermittent mechanical traction plus conventional physical therapy. Participants would undergo 30 minutes of "mechanical traction (with 10-second pull and 5-second rest)" 3 times weekly day after day for four weeks for a total of 12 sessions.
  Interventions: Device: shock waves therapy
- Group (C): (Control group) 20 patients would underwent conventional physical therapy: 3-Group (C): (Control group) 20 patients would underwent conventional physical therapy consisted of "hyperthermia using hot packs (20 minutes), ultrasound (5 minutes), and electrotherapy using TENS (15 minutes) in addition to stretching exercises for the back, iliopsoas, and hamstring muscles and strengthening exercises for the abdominal muscles for 30 minutes".
  Interventions: Device: shock waves therapy

INTERVENTIONS:
Device: shock waves therapy — Group (A): 20 patients would undergo shock waves plus traditional physical therapy. One thousand shock waves (7 times per sec) were applied at 2.5 Hz at low energy flux densities of 0.01-0.16 mJ/mm2 using a 17 mm head 2-Group (B): 20 patients would undergo intermittent mechanical traction plus conventional physical therapy. Participants would undergo 30 minutes of "mechanical traction (with 10-second pull and 5-second rest)"
  Other Names: intermittent mechanical traction

SUMMARY:
investigate the effect of shock wave therapy versus mechanical traction on mechanical low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a common condition that causes tremendous health and socio-economic problems. CLBP is a widespread problem. About 70%-80% of adults in the general population are expected to suffer at least a low back pain episode at some time in their lives1. CLBP is the leading cause of absenteeism at work and creates restrictions on movements, lasting disabilities, and impaired quality of life. Non-specific low back pain is described as low back discomfort, which cannot be attributed to a distinct, known etiology "(e.g., infection, tumors, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome)" 2. Non-specific low back pain is a mechanical musculoskeletal pain that has a symptom that varies according to the physical activity nature 3.

The practice of sitting with a healthy posture and preventing a protracted-standing position can often prevent simple low back pain. However, many kinds of low back pain are addressed with therapies as numerous as the causes of low back pain. The most important treatments are therapeutic measures, such as bed rest, assistive aids, traction therapy, heat, electrical stimulation, and manual therapy are the first choice treatments4. If these methods fails, invasive therapy procedures like nerve roots blocks and epidural injections are employed, and operations are carried out when no reaction to other treatments has been seen or if the disease status is critical. New conservative therapies, including extracorporeal shock wave therapy (ESWT), have recently been embraced 5.

ELIGIBILITY:
Inclusion Criteria:

* Age between (20 and 35 years)
* all subjects suffered from mechanical low back pain

Exclusion Criteria:

* Rheumatoid arthritis or backbone pathologies, and past lumbar vertebrae surgery or cancer were reported

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty Patients between 20 and 35 years of both genders (male and female); all subjects suffered from mechanical low back pain and were picked from the orthopedic hospital in Sohag University. The study took place from April and August 2021 there. Treatment sessions three times a week for four weeks
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire for pain assessment | 1 hour
  The quality and degree of subjective pain are evaluated. The scale comprises 4 subscales examining the sensory, affective, assessment, and other components of pain, pain-intensity responses, and a 5point scale (Present Pain Intensity)

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) | 1 hour
  is a reliable, valid tool for LBP dysfunction assessment. It is one of the more often used measures to evaluate LBP patients' functional state. The RMDQ comprises 24 elements in the LBP-adapted Sickness Impact Profile. The questionnaire was scored by summing the number of 'yes' ranged from 0 (no disability) to 24, were added to the questionnaire (severe disabilities) 12.

OTHER OUTCOMES:
Back Range (BROM) | 1 hour
  instrument is a reliable , objective approach for measuring LBR in all levels regardless of thoracic or hip movement

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abd El Rahim, Sohag, Egypt

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Chung TS, Yang HE, Ahn SJ, Park JH. Herniated Lumbar Disks: Real-time MR Imaging Evaluation during Continuous Traction. Radiology. 2015 Jun;275(3):755-62. doi: 10.1148/radiol.14141400. Epub 2015 Jan 22. PMID 25611735
- [Background] Lee S, Lee D, Park J. Effects of extracorporeal shockwave therapy on patients with chronic low back pain and their dynamic balance ability. J Phys Ther Sci. 2014 Jan;26(1):7-10. doi: 10.1589/jpts.26.7. Epub 2014 Feb 6. PMID 24567665
- [Background] Han H, Lee D, Lee S, Jeon C, Kim T. The effects of extracorporeal shock wave therapy on pain, disability, and depression of chronic low back pain patients. J Phys Ther Sci. 2015 Feb;27(2):397-9. doi: 10.1589/jpts.27.397. Epub 2015 Feb 17. PMID 25729177